CLINICAL TRIAL: NCT03784638
Title: Comparison of Two Different Flap Designs for Bilateral Impacted Mandibular Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Dilek Menziletoglu, Principal Investigator, Konya Necmettin Erbakan Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KonyaNEU
Record Dates: First submitted 2018-12-14; First posted 2018-12-24 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2018-09

CONDITIONS: Impacted Third Molar Tooth
Keywords: trismus; pain; edema; flap design
MeSH Terms: conditions — Trismus; Pain; Edema

STUDY DESIGN:
Intervention Model Description: lingually-based triangle flap design buccaly-based triangular flap design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lingually-based triangle flap design (Experimental): In the experimental group, an incision will be made adjacent to the distal surface of the mandibular second molar, and extended along the sulcus to the distobuccal corner of the mandibular second molar. An oblique vestibular incision will made and extended into the vestibular fornix of the mandible, aligned with the mesiobuccal cusp of the second molar. It was continued posterosuperiorly towards the anterior border of mandibular ramus. The lingually-based triangle flap design will be used.
  Interventions: Procedure: lingually-based triangle flap design
- buccally based triangle flap design (Placebo Comparator): In the control group, an incision will be made from the anterior border of the mandibular second molar. It will be extended along the sulcus to the distobuccal corner of the second molar crown. The incision will be continuous with vertical incision. The buccally based triangle flap design will be used.
  Interventions: Other: buccally based triangular flap design

INTERVENTIONS:
Procedure: lingually-based triangle flap design — A mucoperiosteal lingually-based triangle flap will be raised, a conventional rotary handpiece will be used under irrigation for removing the third molar.Primary wound closure will be accomplished using 4-0 silk sutures. The patients will be invited after one week for removing the sutures.
  Arms: lingually-based triangle flap design
Other: buccally based triangular flap design — A mucoperiosteal buccally based triangular flap will be raised, a conventional rotary handpiece will be used under irrigation for removing the third molar.Primary wound closure will be accomplished using 4-0 silk sutures. The patients will be invited after one week for removing the sutures.
  Arms: buccally based triangle flap design

SUMMARY:
The aim of this study was to compare the effects of lingually-based triangle flap design and buccally based triangular flap design on postoperative swelling, trismus pain after mandibular third molar surgery.

DETAILED DESCRIPTION:
Investigators planned a prospective and split mouth study. Thirty patients is randomly selected. Inclusion criteria is being older than 18 of age, having asymptomatic bilateral mesioangular impacted mandibular third molar (Pell and Gregory class II, position B) fully covered with mucosa and bone, and being otherwise medically healthy. Exclusion criteria is as follows: Alcohol abuse, smoking, pregnancy and acute severe periodontitis.

All surgeries will be carried out by the same surgeon. For each patient, the impacted teeth will be extracted in two sessions using the two different flap design.One side of the patients was selected and labeled as "experimental group". In this group, investigators will use lingually-based triangle flap design while investigators extract the impacted third molar teeth. Other side was accepted as "control group" and in this group, investigators will use buccally based triangular flap design.

In the experimental group, an incision was made adjacent to the distal surface of the mandibular second molar, and extended along the sulcus to the distobuccal corner of the mandibular second molar. An oblique vestibular incision was made and extended into the vestibular fornix of the mandible, aligned with the mesiobuccal cusp of the second molar. It was continued posterosuperiorly towards the anterior border of mandibular ramus. In the control group, an incision will be made from the anterior border of the mandibular second molar. It will be extended along the sulcus to the distobuccal corner of the second molar crown. The incision will be continuous with vertical incision.

A mucoperiosteal flap will be raised, a conventional rotary handpiece will be used under irrigation for removing the third molar.Primary wound closure was accomplished using 4-0 silk sutures. The patients will be invited after one week for removing the sutures.

After the surgery, the patients will be prescribed a 5-day course of 100 mg flurbiprofen twice daily, 1 gr amoxicillin twice daily and chlorhexidine gluconate- benzydamine hydrochloride antiseptic mouthwash every 8 h.There will be at least one month between two surgeries.

The duration of each procedure from the start of the incision to the time of last suture placement will be noted.

Patients are recalled on days 2, 7, 14 postoperative pain, facial swelling, maximum mouth opening, wound dehiscence. For the assesment of the pain, pain scale will be used. For the swelling evaluation, measurement will be done from the different three region on the face.

* Tragus-Pogonion
* Tragus-Labial Commissura
* Angulus Mandible-Lateral canthus

Maximum mouth opening will be noted before and after (one week later) the surgery.

ELIGIBILITY:
Inclusion Criteria:

* symmetrically positioned impacted bilateral mandibular third molars (mesioangular)

Exclusion Criteria:

* pericoronal pathology
* use of medications
* poor oral hygiene
* smoking habit
* pregnancy or lactation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
For edema, the distances between Tragus-Pogonion, Tragus-Labial Commissure, Angulus Mandibula-Lateral Canthus will be measured preoperatively, postoperative 2nd day, 7th day and 14th day surgery. | Up to 2 weeks
  The edema measurement will be done preoperatively, postoperative 2nd day, 7th day and 14th day surgery.

SECONDARY OUTCOMES:
For the assesment of the pain, pain scale will be used. | Up to 1 week
  The patients will fill the pain scale every day until the seventh day after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Menziletoglu, DDS, PhD, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Faculty of Dentistry, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No